CLINICAL TRIAL: NCT05013658
Title: Comparison of the Predictions of Endotracheal Tube Cuff Pressure With Pilot Balloon Palpation and the Value Measured by Manometer Among Anaesthesia Residents in Different Education Years in the Department of Anesthesiology and Reanimation
Brief Title: Comparison of the Predictions of ETTcP With Pilot Balloon Palpation Among Anaesthesia Residents in Different Years
Acronym: ETTcP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Tülay Çardaközü, professor Doctor, Kocaeli University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: manometer1
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Endotracheal Tube Cuff Pressure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- junior (Active Comparator): their anesthesia experiences are between 1 months and 1 year,
  Interventions: Behavioral: pressure measurement
- senior (Active Comparator): Their anesthesia experiences are more than 4 years
  Interventions: Behavioral: pressure measurement

INTERVENTIONS:
Behavioral: pressure measurement — pressure measurement with pilot balloon palpation

SUMMARY:
In routine practice, pressure is often attempted to be adjusted by palpation of the cuff pilot balloon of the endotracheal tube. The aim of our study is to investigate the variation of the reliability of the palpation method, which is widely used in cuff pressure measurement in the absence of a manometer, with clinical experience. Our recommendation is to use an accessible manometer if available.

DETAILED DESCRIPTION:
After the patients were premedicated with an appropriate dose of midazolam, anesthesia was induced with propofol, fentanyl and rocuronium. Endotracheal intubation was performed after ensuring appropriate anaesthesia depth for intubation, by relaxation of the jaw and loss of eyelash reflex. We used 7.5 and 8.0 sizes of sterile ETTs are made of polyvinyl chloride and have a high-volume low-pressure cuffed design that conforms to the shape of the trachea. ETTs for female and male patients and before intubation Tracheal tubes (Tyco Healthcare©, Wollerau Switzerland) cuffs were tested for leakage. The researchers were divided into two groups of 20, with anaesthesia residents (anesthesia experience between 1 months and 1 year, Group J) and those with more than 4 years (Group S). The ETT was placed using the conventional intubation technique with a Macintosh laryngoscope after ensuring appropriate anaesthesia depth for intubation, by relaxation of the jaw and loss of eyelash reflex.. It was asked to swell with air up to cmH2O and a 10 ml injector was used for this. Then Direct pressure measurement was achieved by a cuff manometer calibrated in cmH2O, which was attached to the ETT pilot balloon. The participant was not informed about the actual pressure of cuff. Then the air in the cuff was completely evacuated and the same procedure was repeated with the participant from the other group, the agreement of the two groups to the target value of 25 cmH2O was compared. The order of priority among the groups was randomized according to the closed-envelope method. Controlled positive pressure ventilation was started after the measurement.

In cases in which the cuff pressure was above 30 cmH2O or below 20 cmH2O, the pressure was regulated back to normal limits. During the study, patients were in a supine, head and neck neutral position. Anesthesia was maintained as in our routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergo elective operations with general anesthesia.
2. Ages between 18-75
3. ASA I-II-III patients

Exclusion Criteria:

1. Patient refusal
2. Patients with anticipated difficult airway

   - Tempero-mandibular and atlanto-occipitac joint limitation
3. Having ejection fraction less than 35%
4. Peroperative nasogastric tube inserted patients
5. Patients with a history of sore throat, hoarseness, difficulty swallowing before the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
experience difference | four months
  After intubation, first the assistant doctor with 0-1 year training period and then the assistant doctor with 4-5 years training period will be asked to inflate the cuff to approximately 25 cm H2O cuff pressure by palpation, and the pressure will be measured with a manometer and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: TÜLAY ÇARDAKÖZÜ, Principal Investigator — KOCAELİ ÜNİVERSİTESİ
Locations (1):
- Kocaeli Üniversitesi, Kocaeli, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No